CLINICAL TRIAL: NCT05519527
Title: A Phase 1 Study of Safety and Efficacy of an Anti-CD38 Antibody Drug Conjugate (STI-6129) in Patients With Relapsed or Refractory T-Acute Lymphoblastic Leukemia/Lymphoma (T-ALL) or Acute Myeloid Leukemia (AML)
Brief Title: STI-6129 CD38 ADC for the Treatment of Patients With Relapsed or Refractory Systemic ALL Amyloidosis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: 0 patient accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0113; NCI-2022-07295 (Other: NCI-Clinical Trials Registry)
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Refractory T Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (dose escalation) (Experimental): Participants of the first group will receive the lowest dose level. Participants of each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of STI-6129 is found.
  Interventions: Drug: Part 1 (STI-6129); Drug: Part 2 (STI-6129)
- Part 2 (dose expansion) (Experimental): Participants will receive the dose of STI-6129 found in Part 1 of the study.
  Interventions: Drug: Part 1 (STI-6129); Drug: Part 2 (STI-6129)

INTERVENTIONS:
Drug: Part 1 (STI-6129) — Given by vein (IV)
Drug: Part 2 (STI-6129) — Given by vein (IV)

SUMMARY:
This is an open-label, phase 1b/2 trial. It is designed to identify the recommended phase 2 dose (RP2D) of STI-6129, and the safety and efficacy of this anti-CD38-Duostatin 5.2 antibody-drug conjugate (ADC) for the treatment of R/R T-ALL and AML who have exhausted standard of care treatment.

DETAILED DESCRIPTION:
Primary Objective:

* To assess in patients with R/R T-ALL or AML
* Maximum tolerated dose of STI-6129
* Phase 2 recommended dose
* Safety of STI-6129

Secondary Objectives:

* Efficacy of STI-6129, overall response rate (CR+CRi+MLFS)
* Evaluate rate of negative measurable residual disease (MRD)
* Evaluate overall survival, duration of response, event-free survival
* No. of patients transitioning to stem-cell transplantation

Exploratory Objectives:

- Evaluate the association of biomarkers with safety and efficacy in patients with R/R T-ALL or AML treated with STI-6129 CD38 ADC STI-6129 - R/R T-ALL, AML

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in the study, patients must satisfy all inclusion criteria, as follows:

1. Age greater than or equal to 18 years.
2. Confirmed diagnosis of R/R T-ALL or R/R AML by bone marrow evaluation. Note that patients must have failed treatment with available therapies known to be active for treatment of their T-ALL/AML
3. ECOG performance status of 0, 1, or 2
4. Pulse oximetry greater than or equal to 92% on room air
5. Be willing and able to comply with the study schedule and all other protocol requirements
6. Females of childbearing potential (FCBP), defined as a sexually mature woman who has not undergone a hysterectomy or tubal ligation or who has not been naturally postmenopausal for at least 24 consecutive months, must have a negative pregnancy test during the Screening Period prior to treatment. All heterosexually active FCBP and all heterosexually active male patients must agree to use effective methods of birth control throughout the study

Subject Exclusion Criteria:

To be enrolled in the study, patients must not satisfy any of the following exclusion criteria:

1. A diagnosis of other malignancies if the malignancy has required therapy within the last 3 months or is not in complete remission. Exceptions are non-metastatic basal cell or squamous cell carcinomas of the skin or prostate cancer or in situ cancer that does not require further active treatment or is well under control
2. Treatment with an allogeneic hematopoietic stem cell transplantation (HSCT) within 3 months prior to the planned infusion of STI-6129, or active graft-versus-host disease (GVHD) following the allogeneic transplant, or a requirement for currently receiving immunosuppressive therapy following the allogeneic transplant.
3. Must be off calcineurin inhibitors for at least 4 weeks prior to study treatment.
4. New York Heart Association (NYHA) class greater than or equal to 3
5. Left ventricular ejection fraction (LVEF) < 40%.
6. The following baseline chemistry laboratory results at Screening:

   1. Serum creatinine > 2.0 x the upper limit of normal (ULN), or estimated creatinine clearance < 60 mL/min (using the Cockcroft-Gault equation).
   2. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3x the upper limit of normal (ULN) or serum total bilirubin > 1.5x ULN (except for patients in or leukemia involvement)
7. Pregnancy or currently breastfeeding
8. Patients with greater than Grade 3 neuropathy or Grade 2 neuropathy with associated pain
9. Active bacterial, viral, or fungal infection at the time of the infusion of STI-6129; patients with ongoing use of prophylactic antibiotics, antifungal agents, or antiviral agents, or infection controlled on antimicrobial agents remain eligible as long as there is no evidence of active infection
10. Uncontrolled human immunodeficiency virus (HIV) infection, human T-cell leukemia virus type 1 (HTLV1) infection, or active hepatitis B virus (HBV) or hepatitis C virus (HCV) viremia or are at risk for HBV reactivation (at risk for HBV reactivation is defined as being HBs antigen positive, or anti-HBc-antibody positive), or are positive for HBV deoxyribonucleic acid (DNA). HCV ribonucleic acid (RNA) must be undetectable by laboratory test.
11. Have a prolongation in QTcF (Fridericia correction formula) > 480 msec on a baseline ECG
12. Any condition including the presence of laboratory abnormalities that places the patient at an unacceptable risk if the patient was to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Severity of the adverse events (Aes) -The severity of the adverse events (Aes) will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) V.5 | through completion of study or an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Maiti, MBBS, Principal Investigator — amaiti@mdanderson.org

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org